CLINICAL TRIAL: NCT00667043
Title: Remifentanil and Propofol Versus Fentanyl and Midazolam for Sedation During Therapeutic Hypothermia. A Randomised, Controlled Trial
Acronym: Cool Sedation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OPI 07 001
Record Dates: First submitted 2008-04-23; First posted 2008-04-25 (Estimated); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Hypothermia
Keywords: therapeutic hypothermia; cardiac arrest; sedation; remifentanil; propofol; fentanyl; midazolam
MeSH Terms: conditions — Hypothermia; Heart Arrest | interventions — Remifentanil; Propofol; Fentanyl; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study group 1 (Active Comparator): Midazolam and fentanyl; continuous intravenous infusions
  Interventions: Drug: fentanyl and midazolam
- Study group 2 (Active Comparator): Propofol and remifentanil; continuous intravenous infusion
  Interventions: Drug: remifentanil and propofol

INTERVENTIONS:
Drug: remifentanil and propofol — Patients will receive: propofol, continuous intravenous infusion, concentration 10 mg/ml, 1-4 mg/kg/hour and remifentanil; continuous intravenous infusion 0,050 mg/ml, 0.1-0.3 microgram/kg/min. Drugs are administered to sedate the patients as part of normal treatment for as long as sedation is needed. Doses are titrated to achieve the desired level of sedation.
  Arms: Study group 2
Drug: fentanyl and midazolam — Patients will receive: midazolam; continuous intravenous infusion, concentration 5 mg/ml, 2-10 mg/hour and fentanyl; continuous intravenous infusion, concentration 0,050 mg/ml, 0.025-0.5 mg/hour. Drugs are administered to sedate the patients as part of normal treatment for as long as sedation is needed. Doses are titrated to achieve the desired level of sedation.
  Arms: Study group 1

SUMMARY:
The aim of this study is to increase knowledge about drug properties and effects during therapeutic hypothermia. The primary end point of this study is the time from termination of sedation to extubation in patients treated with therapeutic hypothermia, after treatment with the combination remifentanil and propofol versus that of fentanyl and midazolam.

ELIGIBILITY:
Inclusion Criteria:

* Treatment with therapeutic hypothermia following cardiac arrest (33-34°C) and analgesia/sedation required
* Patients must be 18 years or older
* Inclusion must be approved by the attending physician

Exclusion Criteria:

* Pregnant women
* Cardiovascular unstable patients in a deteriorating circulatory status which require multiple other therapeutic measures that makes participation practically impossible
* Liver or renal failure defined as sequential organ failure assessment (SOFA)-score 3 or 4
* History of drug allergies, or contraindications for the study drugs
* Patients using a scheduled dose of any of the study drugs.
* Patients with a known substance abuse of opioids or benzodiazepines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-04; Primary Completion 2009-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
time from termination of sedation to extubation in patients treated with therapeutic hypothermia, after treatment with the combination remifentanil and propofol versus that of fentanyl and midazolam. | 2010

CONTACTS AND LOCATIONS:
Overall Officials: Pål Klepstad, MD, PhD, Study Director — National Taiwan Normal University
Locations (2):
- Norway (2):
  - Stavanger University Hospital, Stavanger, Rogaland
  - St. Olavs Hospital, Trondheim, Sør-Trøndelag

REFERENCES:
- [Result] Bjelland TW, Dale O, Kaisen K, Haugen BO, Lydersen S, Strand K, Klepstad P. Propofol and remifentanil versus midazolam and fentanyl for sedation during therapeutic hypothermia after cardiac arrest: a randomised trial. Intensive Care Med. 2012 Jun;38(6):959-67. doi: 10.1007/s00134-012-2540-1. Epub 2012 Apr 12. PMID 22527063